CLINICAL TRIAL: NCT02228525
Title: A Phase II Study of the Selective Inhibitor of Nuclear Export (SINE) Selinexor (KPT-330) in Patients With Myelodysplastic Syndromes
Brief Title: Selective Inhibitor of Nuclear Export (SINE) Selinexor (KPT-330) in Patients With Myelodysplastic Syndromes
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: M.D. Anderson Cancer Center (Other); Columbia University (Other); Karyopharm Therapeutics Inc (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 14-005
Record Dates: First submitted 2014-08-27; First posted 2014-08-29 (Estimated); Results first posted 2022-03-09 (Actual); Last update posted 2022-03-09 (Actual); Status verified 2021-04

CONDITIONS: Myelodysplastic Syndromes
Keywords: Selinexor (KPT-330); Selective Inhibitor of Nuclear Export (SINE); 14-005
MeSH Terms: conditions — Myelodysplastic Syndromes | interventions — selinexor

ARMS (1):
- selinexor (KPT-330) (Experimental): Patients with myelodysplastic syndromes who are refractory to hypomethylating agents (decitabine or 5-azacytidine) will receive oral selinexor at a starting dose of 60 mg twice weekly for 2 weeks, followed by 1 week of no therapy. Dose reductions are permitted for patients who are benefiting from selinexor but have poor tolerance. After discontinuation from treatment, patients will be followed by the study staff for survival status approximately every three months.
  Interventions: Drug: selinexor (KPT-330)

INTERVENTIONS:
Drug: selinexor (KPT-330)

SUMMARY:
The purpose of this study is to see if selinexor will improve the blood counts and bone marrow function in people with your type of MDS.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent in accordance with federal, local, and institutional guidelines
* Age ≥18 years
* Patients with Myelodysplastic Syndromes refractory (primary or acquired resistance) to hypomethylating agents(decitabine or 5-azacytidine). At least 4 1- month cycles of prior decitabine or SGI-110 OR 6 1-month cycles of 5-azacytidine (IV, subcutaneous, or oral is required unless the patient has progressive disease prior to completing the required number of cycles.
* Histologically confirmed diagnosis of a Myelodysplastic Syndrome, meeting criteria for any subtype in the FAB or WHO classification systems with any IPSS score.
* Patients with MDS who relapse after allogeneic stem cell transplant are eligible if they received standard dose decitabine or 5-azacytidine prior to or after stem cell transplant as defined in inclusion criteria 3.
* If patient has undergone prior allogeneic stem cell transplant, they must be greater than 100 days post transplant and have ≤ grade 2 graft-versus-host disease
* There is no upper limit on the number of prior treatments provided all inclusion/exclusion criteria are met.
* Eastern Cooperative Oncology Group (ECOG) Performance Status of 0-2
* Patients receiving erythropoietin (darbepoetin, epoetin alfa) must be on a stable dose and with stable transfusion requirement or hemoglobin level during the 8 weeks prior to study entry.
* Adequate hepatic function within 21 days prior to C1D1: total bilirubin <2 times the upper limit of normal (ULN), asparate aminotransferase (AST) <2.5 times ULN and alanine aminotransferase (ALT) <2.5 times ULN.
* Adequate renal function within 21 days prior to C1D1: estimated creatinine clearance of ≥ 30 mL/min, calculated using the formula of Cockcroft and Gault.
* Female patients of child-bearing potential must agree to use dual methods of contraception and have a negative serum pregnancy test at screening, and male patients must use an effective barrier method of contraception if sexually active with a female of child-bearing potential. Acceptable methods of contraception are condoms with contraceptive foam, oral, implantable or injectable contraceptives, contraceptive patch, intrauterine device, diaphragm with spermicidal gel, or a sexual partner who is surgically sterilized or post-menopausal. For both male and female patients, effective methods of contraception must be used throughout the study and for three months following the last dose.

Exclusion Criteria:

* Patients who are pregnant or lactating;
* Chemotherapy or immunotherapy or any other anticancer therapy ≤3 weeks prior to cycle 1 day 1. Hydroxyurea may be continued until 72 hours prior to first dose and at least 24 hours before the baseline bone marrow aspiration is performed;
* Major surgery within four weeks before Day 1;
* Unstable cardiovascular function defined as symptomatic ischemia, uncontrolled clinically significant conduction abnormalities (ie: ventricular tachycardia on antiarrhythmics are excluded and 1st degree AV block or asymptomatic LAFB/RBBB will not be excluded), congestive heart failure (CHF) of NYHA Class ≥3, or myocardial infarction (MI) within 3 months;
* Uncontrolled active infection requiring systemic antibiotics, antivirals, or antifungals within one week prior to first dose; Prophylactic antimicrobials are permitted.
* Known to be HIV seropositive;
* Known active hepatitis A, B, or C infection; or known to be positive for HCV RNA or HBsAg (HBV surface antigen);
* Patients with another active malignancy. Asymptomatic sites of disease are not considered active. Treated or untreated sites of disease may be considered inactive if they are stable for at least 2 months and are not expected to require therapy for 4 months.
* Patients with significantly diseased or obstructed gastrointestinal tract or uncontrolled vomiting or diarrhea.
* Grade ≥2 peripheral neuropathy at baseline (within 21 days prior to cycle 1 day 1).
* History of seizures, movement disorders or cerebrovascular accident within the past 1 years prior to cycle 1 day 1.
* Patients with macular degeneration with markedly decreased visual acuity, patients with markedly decreased visual acuity (no specific etiology) or uncontrolled glaucoma.
* Patients who are significantly below their ideal body weight (BMI < 17)..
* Serious psychiatric or medical conditions that could interfere with treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2014-08-27 (Actual); Primary Completion 2021-04-06 (Actual); Study Completion 2021-04-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Virginia Klimek, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan Kettering Cancer Center, New York, New York, United States

REFERENCES:
- [Derived] Taylor J, Mi X, Penson AV, Paffenholz SV, Alvarez K, Sigler A, Chung SS, Rampal RK, Park JH, Stein EM, Tallman MS, Sen F, Gonen M, Abdel-Wahab O, Klimek VM. Safety and activity of selinexor in patients with myelodysplastic syndromes or oligoblastic acute myeloid leukaemia refractory to hypomethylating agents: a single-centre, single-arm, phase 2 trial. Lancet Haematol. 2020 Aug;7(8):e566-e574. doi: 10.1016/S2352-3026(20)30209-X. PMID 32735836
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org/

RESULTS

PARTICIPANT FLOW:
Groups:
- Selinexor (KPT-330): Patients with myelodysplastic syndromes who are refractory to hypomethylating agents (decitabine or 5-azacytidine) will receive oral selinexor at a starting dose of 60 mg twice weekly for 2 weeks, followed by 1 week of no therapy. Dose reductions are permitted for patients who are benefiting from selinexor but have poor tolerance. After discontinuation from treatment, patients will be followed by the study staff for survival status approximately every three months.
  selinexor (KPT-330)
Period: Overall Study
Arm/Group | Selinexor (KPT-330)
Started | 25
Completed | 25
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Selinexor (KPT-330)
Number analyzed (Participants) | 25
Age, Continuous [Median (Full Range); unit: years] | 77 [70 to 81]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 21
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 8
  Unknown or Not Reported | 17
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 23
  More than one race | 0
  Unknown or Not Reported | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 25

OUTCOME MEASURES:

1. Primary Outcome: Best Overall Response Rate
Description: Using a Simon's two-stage minimax design, this trial will accrue a maximum of 20 patients. Early termination may occur if no responses are observed in the first 13 patients. If at least one response is observed, the trial will continue to the maximum sample size. At the end of the trial, the treatment strategy will be considered promising in this patient population if at least 3 patients achieve a response. The type I and type II errors are set at 0.10.
Time Frame: 2 years
Measure: Number (95% Confidence Interval); unit: Percentage of participants with response
Arm/Group | Selinexor (KPT-330)
Number analyzed (Participants) | 25
Percentage of participants with response | 26 [10 to 48]

2. Secondary Outcome: Response Duration
Description: Response duration will be calculated among patients who achieve a response of HI, mCR, PR or CR using Kaplan-Meier methodology. Median duration of response and the corresponding 95% confidence interval will be estimated.
Time Frame: 2 years
Measure: Median (Full Range); unit: months
Arm/Group | Selinexor (KPT-330)
Number analyzed (Participants) | 25
months | 6.3 [2.1 to 7.8]

3. Secondary Outcome: Overall Survival
Description: Overall survival from the time of study enrollment will be calculated using Kaplan-Meier methodology. Overall survival curves will be displayed for the study population along with selected quantiles and corresponding 95% confidence intervals of survival.
Time Frame: 2 years
Measure: Median (Full Range); unit: months
Arm/Group | Selinexor (KPT-330)
Number analyzed (Participants) | 25
months | 8.5 [6.7 to 12.2]

4. Secondary Outcome: Participants Evaluated for Adverse Events
Description: The safety and tolerability of Selinexor and ST will be evaluated by means of drug related AE reports, physical examinations, and laboratory safety evaluations. Common Terminology Criteria for Adverse Events (CTCAE) V4.03 will be used for grading of AEs.
Time Frame: 2 years
Measure: Count of Participants; unit: Participants
Arm/Group | Selinexor (KPT-330)
Number analyzed (Participants) | 25
Participants | 25

ADVERSE EVENTS:
Time Frame: 2 years
Arm/Group | Selinexor (KPT-330)
All-Cause Mortality (participants affected / at risk) | 7/25
Serious Adverse Events (participants affected / at risk) | 0/25
Other Adverse Events (participants affected / at risk) | 25/25
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Selinexor (KPT-330) (N=25)
Anorexia or weight loss (Metabolism and nutrition disorders) | 10
Fatigue (General disorders) | 14
Malaise (General disorders) | 2
Diarrhea (Gastrointestinal disorders) | 5
Dysgeusia (Nervous system disorders) | 4
Increased alanine aminotransferase (Investigations) | 2
Hyperglycaemia (Metabolism and nutrition disorders) | 9
Hyperkalaemia (Metabolism and nutrition disorders) | 2
Hypoalbuminaemia (Metabolism and nutrition disorders) | 6
Hypocalcaemia (Metabolism and nutrition disorders) | 3
Hyponatraemia (Metabolism and nutrition disorders) | 11
Nausea or vomiting (Gastrointestinal disorders) | 14
Decreased white blood cell count (Investigations) | 4
Decreased neutrophil count (Investigations) | 7
Febrile neutropenia (Blood and lymphatic system disorders) | 2
Anaemia (Blood and lymphatic system disorders) | 3
Decreased platelet count (Investigations) | 12

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-01-25): https://cdn.clinicaltrials.gov/large-docs/25/NCT02228525/Prot_SAP_000.pdf